CLINICAL TRIAL: NCT03539055
Title: Efficacy of Short Term Dabigatran Etexilate Followed by Aspirin Monotherapy After LAA (Left Atrial Appendage) Device Closure (the DEA-LAA Study).
Acronym: DEA-LAA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Arvindh Kanagasundram, Assistant Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DEA-LAA
Record Dates: First submitted 2018-05-12; First posted 2018-05-29 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation; Device Related Thrombus; Left Atrial Appendage Thrombosis; Watchman LAA Closure Device
Keywords: DRT; Device related thrombus; Dabigatran etexilate; Aspirin; Watchman
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran

STUDY DESIGN:
Intervention Model Description: Prospective single arm intervention of dabigatran etexilate with aspirin for 90 days following Watchman LAA device closure to prevent device related thrombus (DRT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Dabigatran 75 or 150mg BID x 90 days plus ASA 81mg daily.
  Single arm, prospective unblinded study on post Watchman LAA closure device implant anti-coagulation management at a primary center (Vanderbilt Medical Center) and up to 5 additional high volume LAA implant centers. This trial will be designed to evaluate the use of dabigatran for 90 days post implantation of an LAA closure device (Watchman LAA Closure Device, Boston Scientific Inc.)
  Interventions: Drug: Dabigatran Etexilate Oral Capsule

INTERVENTIONS:
Drug: Dabigatran Etexilate Oral Capsule — Oral use of Dabigatran etexilate for 90 days BID per product labeling for dosage to reduce incidence of device related thrombus after implantation of a Watchman LAA device.
  Other Names: Pradaxa

SUMMARY:
Single arm, prospective unblinded study on post Watchman LAA closure device implant anti-coagulation management at a primary center (Vanderbilt Medical Center) and up to 5 additional high volume LAA implant centers. This trial will be designed to evaluate the use of dabigatran for 90 days post implantation of an LAA closure device (Watchman LAA Closure Device, Boston Scientific Inc.) to prevent device related thrombus.

DETAILED DESCRIPTION:
Single arm, prospective unblinded study on post Watchman LAA closure device implant anti-coagulation management at a primary center (Vanderbilt Medical Center) and up to 5 additional high volume LAA implant centers. This trial will be designed to evaluate the use of dabigatran for 90 days post implantation of an LAA closure device (Watchman LAA Closure Device, Boston Scientific Inc.).

The drug will be initiated on the morning following device implantation, taken BID per package insert dosing and until follow-up 90-day post implant TEE. Aspirin monotherapy will be utilized in conjunction at 81 mg for up to 12 months, after which the patients will be exited from the study and further treatment decisions will be made by the following physician (see Schedule of Study Procedures at end of protocol). The objective of this trial is to evaluate safety and efficacy of a 90-day period of dabigatran etexilate following LAA closure to prevent device associated thrombus, while minimizing adverse bleeding by eliminating the need for clopidogrel.

This is a single arm pilot study with the option (pending collaboration with additional funding source) to expand to a full single arm non-inferiority trial design with 80% power to detect a 1.4% difference with the non-inferiority margin 1% in absolute rate of DAT (control rate 3.9%).

Prospective, non-randomized single arm study. Comparison will be made to historical controls based on published one year DAT rates from PROTECT-AF, PREVAIL clinical trials, and EWOLUTION, and ACP/Amulet registries.

Echocardiography (TEE) will be performed at 90 days (3 months, +/- 2-week window), and again at 1-year post implant (+/- 4 weeks). Selected images will be interpreted by echo lab at coordinating center in an anonymous fashion (patient data de-identified). Ideal imaging will incorporate 0, 45, 90 and 135 degree angled views on the device at follow up.

Drug will be dispensed as part of the clinical trial supplied from the sponsor and each patient will receive a complete 90 days' supply up front. They will have a drug visit on the day of TEE with the research coordinator to hand back any remaining dabigatran, with clear instruction to stop the drug and only take ASA following confirmation of closure on TEE (no peri-device leak on Doppler of >5mm). A decision to continue anti-coagulation post closure 90day TEE will be made by the physician discretion based on TEE findings. If thrombus is found at the 90 days TEE, anti-coagulation may be extended another 6 weeks with repeat TEE imaging to confirm clot resolution at the discretion of the investigator. In the unlikely event of embolization or Doppler leak >5mm, decision on extending anti-coagulation, or re-implanting a device will be made by the following physician.

Additional baseline data collection: Patient demographics, medical history, age, sex, and prior use of anti-coagulants or anti-platelet medications will be collected. CHADS 2 Vasc, and HAS-BLED score calculated. Main indication for LAA closure must be documented. Baseline CBC and BMP required on day of implant or up to 1 week pre-procedure (typical standard of care labs at time of implant). This will include a recent calculation of Creatinine Clearance (using Cockroft Gault and using patients actual body weight) and dosing of study drug will be made in accordance (see below). Repeat PCV or hematocrit on the morning after Watchman LAAC implantation will be per hospital standard. PCV or hematocrit value pre-implant and at the post 90-day visit will be analyzed.

Calculation for dabigatran dosing:

CCr={ (l40-age) x weight in kg)/(72 x SCr) } x 0.85 (if female)

Implant procedure variables to collect include access site, sheath used for deployment (WAS), device size at implant and number of implant attempts. LA pressure mean if available. Presence of angiography contrast or Doppler Echo leak, thrombus, or pericardial effusion post implant will be recorded. At 90 days, TEE report findings and image review (standard of care) with drug dosing visit with research coordinator and return of any remaining study drug.

1 year TEE (standard of care) with a research exit visit with MD, physician extender, or research coordinator, with documentation of ASA tolerance, dosing, and any late bleeding episodes or hospitalizations (typically should be reported as AE/SAE when first knowledge of event is determined). TEE images will be sent to the primary study site (Vanderbilt University Medical Center) and core TEE lab will review to confirm presence or absence of DAT. In cases of CTA utilized for follow up, similarly images will be reviewed by chest radiology team at Vanderbilt.

Medication administration with 90 days of dabigatran to be dispensed by pharmacy ideally one time (180 capsules).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female sex, age >18 years.
2. CHADS2 Vascular score of 3-9 and HAS BLED score 2 or higher meeting CMS coverage criteria for Watchman LAA closure device implantation.
3. Able to give informed consent.
4. Life expectancy of > 1year in the judgment of the implanting physician and shared decision-making physician.

Exclusion Criteria:

1. Unable to give informed consent
2. History of confirmed allergy to dabigatran etexilate
3. Active cerebral bleeding, or active non-cerebral bleeding requiring blood transfusions (any absolute contra-indications to anti-coagulation).
4. History of intraocular, spinal, retroperitoneal or a traumatic intra-articular bleeding unless the causative factor has been permanently eliminated or repaired (e.g. by surgery)
5. Gastrointestinal (GI) haemorrhage within one month prior to screening, unless, in the opinion of the Investigator, the cause has been permanently eliminated (e.g. by surgery)
6. Major bleeding episode (reduction in the haemoglobin level of at least 2g/dL, transfusion of at least two units of blood, or symptomatic bleeding in a critical area or organ) including life-threatening bleeding episode (symptomatic intracranial bleeding, bleeding with a decrease in the haemoglobin level of at least 5g/dL or bleeding requiring transfusion of at least 4 units of blood or inotropic agents or necessitating surgery) in one month prior to screening visit
7. Intolerance to dabigatran, if medication naïve, or other contra-indications as per the USPI, including ESRD on hemodialysis or GFR < 15ml/min, or concomitant use of rifampin.
8. History of non-compliance, inability to follow-up.
9. Pre-menopausal women (last menstruation ≤ 1 year prior to screening) who are not surgically sterile.
10. Ischemic stroke or hemorrhagic stroke within 90 days of LAA placement.
11. Anatomy unsuitable for LAA closure (incomplete surgical LAA ligation without suitable anatomy for Watchman placement. LAA ostial measurements >31mm, or <17mm in all views).
12. Requires long-term oral anticoagulation therapy for a condition other than atrial fibrillation.
13. ASA allergy, or confirmed allergy to nickel.
14. Prior PFO or ASD closure device or prosthetic or mechanical heart valve.
15. Acute MI within 90 days.
16. Platelets <50,000 at time of Watchman LAAC implantation.
17. Active endocarditis.
18. Planning for endocardial catheter AF or left atrial ablation within 90 days of Watchman implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arvindh N Kanagasundram, MD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
RedCap database, central to primary center, online, web based and HIPAA compliant. Password protected and encrypted database.

REFERENCES:
- [Background] Aryana A, Singh SK, Singh SM, O'Neill PG, Bowers MR, Allen SL, Lewandowski SL, Vierra EC, d'Avila A. Association between incomplete surgical ligation of left atrial appendage and stroke and systemic embolization. Heart Rhythm. 2015 Jul;12(7):1431-7. doi: 10.1016/j.hrthm.2015.03.028. Epub 2015 May 18. PMID 25998141
- [Background] Lim YM, Kim JS, Kim TH, Uhm JS, Shim CY, Joung B, Hong GR, Lee MH, Jang YS, Pak HN. Delayed left atrial appendage contrast filling in computed tomograms after percutaneous left atrial appendage occlusion. J Cardiol. 2017 Dec;70(6):571-577. doi: 10.1016/j.jjcc.2017.04.007. Epub 2017 May 22. PMID 28546017
- [Background] Kaneko H, Neuss M, Weissenborn J, Butter C. Predictors of thrombus formation after percutaneous left atrial appendage closure using the WATCHMAN device. Heart Vessels. 2017 Sep;32(9):1137-1143. doi: 10.1007/s00380-017-0971-x. Epub 2017 May 5. PMID 28477098
- [Background] Fauchier L, Cinaud A, Brigadeau F, Lepillier A, Pierre B, Abbey S, Fatemi M, Franceschi F, Guedeney P, Jacon P, Paziaud O, Venier S, Deharo JC, Gras D, Klug D, Mansourati J, Montalescot G, Piot O, Defaye P. Device-Related Thrombosis After Percutaneous Left Atrial Appendage Occlusion for Atrial Fibrillation. J Am Coll Cardiol. 2018 Apr 10;71(14):1528-1536. doi: 10.1016/j.jacc.2018.01.076. PMID 29622159
- [Background] Pracon R, Bangalore S, Dzielinska Z, Konka M, Kepka C, Kruk M, Kaczmarska-Dyrda E, Petryka-Mazurkiewicz J, Bujak S, Solecki M, Pskit A, Dabrowska A, Sieradzki B, Plonski A, Ruzyllo W, Witkowski A, Demkow M. Device Thrombosis After Percutaneous Left Atrial Appendage Occlusion Is Related to Patient and Procedural Characteristics but Not to Duration of Postimplantation Dual Antiplatelet Therapy. Circ Cardiovasc Interv. 2018 Mar;11(3):e005997. doi: 10.1161/CIRCINTERVENTIONS.117.005997. PMID 29463510
- [Background] Bergmann MW, Ince H, Kische S, Schmitz T, Meincke F, Schmidt B, Foley D, Betts TR, Grygier M, Protopopov AV, Stein KM, Boersma LVA. Real-world safety and efficacy of WATCHMAN LAA closure at one year in patients on dual antiplatelet therapy: results of the DAPT subgroup from the EWOLUTION all-comers study. EuroIntervention. 2018 Apr 20;13(17):2003-2011. doi: 10.4244/EIJ-D-17-00672. PMID 29313819

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: Dabigatran 75 or 150mg BID x 90 days plus ASA 81mg daily.
  Single arm, prospective unblinded study on post Watchman LAA closure device implant anti-coagulation management at a primary center (Vanderbilt Medical Center) and up to 5 additional high volume LAA implant centers. This trial will be designed to evaluate the use of dabigatran for 90 days post implantation of an LAA closure device (Watchman LAA Closure Device, Boston Scientific Inc.)
  Dabigatran Etexilate Oral Capsule: Oral use of Dabigatran etexilate for 90 days BID per product labeling for dosage to reduce incidence of device related thrombus after implantation of a Watchman LAA device.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 100
Completed | 84
Not Completed | 16
Not completed — Death | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Screen Fail | 7
Not completed — Drug Intolerance | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.41 (7.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 63
  Sex: Female | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 94
  More than one race | 0
  Unknown or Not Reported | 0
CHADS2 Vascular Score [Median (Standard Deviation); unit: percentage] — CHADS2 score was assessed by combining score of 5 risk factors (congestive heart failure history, hypertension history, age >=75 years, diabetes mellitus history and stroke/transient ischemic attack symptoms previously). Total CHADS2 score ranged from 0-5 where 0 =low risk and 5 =high risk of stroke.
  percentage | 4.3 (1.3)
HAS-BLED Score [Mean (Standard Deviation); unit: percentage] — HAS-BLED scoring scale was used to estimate the risk of bleeding. HAS-BLED score was calculated based on 9 risk factors (hypertension, renal disease, liver disease, stroke history, prior major bleeding or predisposition to bleeding, labile international normalized ratio (INR), age >65 years, medication usage predisposing to bleeding and alcohol use). Total HAS-BLED score ranged from 0 to 9 where 0 = low risk and >=3 = high risk of bleed.
  percentage | 3.5 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Device Related Thrombus (DRT) at 90 Days
Description: Transesophageal echocardiogram or CT angiography determined presence of DRT at 90 days
Time Frame: Baseline to 90 days
Population: • Withdrawal from study (up to 90 days)
  1. Failed to meet inclusion/exclusion criteria (n=5)
  2. Withdrew consent (n=2)
  3. Unable to complete and initiate 90 days or dabigatran (n=2)
  4. Death prior to 90-day TEE follow-up (n=1)
  5. Coud not get 90 day TEE (n=2)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 88
Participants | 1

2. Primary Outcome: Device Related Thrombus (DRT) at 1 Year
Description: Transesophageal echocardiogram or CT angiography determined presence of DRT at 1 year post implant
Time Frame: 90 days to 1 year
Population: • Withdrawal from study (90days to 1 year )
  1. Covid delay for 12 month TEE (n=5)
  2. Patient death between 90 days and 1 year TEE (n=2_
  3. Health decline with inability to get TEE (n=1)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 80
Participants | 0

3. Secondary Outcome: Includes Ischemic Stroke, Peripheral Thrombo-embolic Events and Major Bleeding Events
Description: Ischemic stroke, peripheral thrombo-embolic events and major bleeding events on dabigatran etexilate at 90 days
Time Frame: Baseline to 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 88
Participants
  Ischemic Stroke | 0
  Peripheral thrombo-embolic events | 0
  Major Bleeds requiring intervention | 3

ADVERSE EVENTS:
Time Frame: Enrollment to one year post procedure
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 4/88
Serious Adverse Events (participants affected / at risk) | 8/88
Other Adverse Events (participants affected / at risk) | 11/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=88)
GI Bleeding (Gastrointestinal disorders) | 6 — GI Bleeding requiring transfusion
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 — Respiratory failure requiring admission
Pericardial effusion (Cardiac disorders) | 1 — Pericardial effusion requiring intervention
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=88)
Gastrointestinal side effect (Gastrointestinal disorders) | 4 — GI irritation (without major bleeding)
Non-ST elevation MI (Cardiac disorders) | 1 — Minor cardiac event
Blurred Vision (Eye disorders) | 1
Pericardial Pain (Cardiac disorders) | 1
Pulmonary infection (Respiratory, thoracic and mediastinal disorders) | 1
Headache (General disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 — Exacerbation of rheumatic arthritis symptoms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT03539055/Prot_SAP_000.pdf